CLINICAL TRIAL: NCT04544891
Title: Prognostic Significance of the TREM-1 Pathway Activation in COVID-19
Brief Title: TREM-1 Pathway Activation in COVID-19
Acronym: CoviTrem1
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Limoges (Other); Inotrem (Industry)
Responsible Party: Principal Investigator, Gibot Sébastien, Pr, Central Hospital, Nancy, France
Other Study IDs: 2020PI120
Record Dates: First submitted 2020-09-09; First posted 2020-09-10 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — Blood will be collected every 3 days until Day 28, discharge, or death

SUMMARY:
Severe Acute Respiratory Syndrome-Corona Virus-2 infection results in a mild infection in most of the patients. However, 15-20% require hospitalization, and among them, 15-20% will develop acute respiratory failure, leading to their admission in Intensive Care Unit. There are no accepted predictive criteria for aggravation. Severe forms of Coronavirus induced disease-19 (COVID-19) are the consequence of endotheliopathy, and hyperinflammatory and pro-coagulant state. The Triggering Receptor Expressed on Myeloid cells-1 (TREM-1) is an immunoreceptor that acts as an amplifier of the inflammatory response. TREM-1 is expressed on myeloid and endothelial cells. Its activation leads to endothelial activation and damage, hyperinflammatory, and pro-coagulant state. TREM-1 activation is associated with poor outcome during septic shock and myocardial infarction.

We here aim at investigating the relationship between TREM-1 pathway activation and clinical degradation and outcome of COVID-19 hospitalized patients.

ELIGIBILITY:
Inclusion Criteria Consecutive COVID-19 hospitalized patients for less than 3 days

Exclusion Criteria:

No consent Pregnancy protected populations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1000 consecutive COVID-19 patients hospitalized for less than 3 days; among them at least 200 patients hospitalized in ICU (primary admission or secondary transfer from the ward)
Sampling Method: Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
prognostic value of the TREM-1 pathway activation on clinical worsening | day 28

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU Limoges, Limoges
  - Central hospital, Nancy

IPD SHARING:
Plan to Share IPD: Undecided